CLINICAL TRIAL: NCT04366388
Title: Assessing a New Tool to Assess Frailty in Frail Hospitalized Elderly
Status: Enrolling by invitation | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kenneth Madden, Principal Investigator, University of British Columbia
Other Study IDs: H19-04017
Record Dates: First submitted 2020-04-15; First posted 2020-04-28 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Frail Elderly Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Frail hospitalized old adults: Over than 65-years of age Admitted into Acute Unit Nonambulatory
  Interventions: Device: ActivPAL3 VT (PAL Technologies Ltd).

INTERVENTIONS:
Device: ActivPAL3 VT (PAL Technologies Ltd). — . The ActivPAL will be fitted by a trained research assistant on the mid-thigh of the participants' dominant leg. ActivPALs have an inclinometer that detects the joint angle of the thigh to capture lying, sitting, standing, and stepping activities.
  Other Names: ActivPal sensor

SUMMARY:
The major purpose of this study is to establish the use of daily step counts as inexpensive, easy to measure marker for frailty and sarcopenia in an inpatient population of older adults.

DETAILED DESCRIPTION:
The total time involved to complete study procedures will be between 2-3 hours at your enrollment and up to 10 minutes at your discharge. Investigators will invite participants to enrol in this study at your admission and discharge days.

Firstly, Investigators would like to collect some demographic data, including participants age and gender.

Then Investigators will ask participants to check their blood pressure and heart rate, weight, height and Body Mass Index.

Also Investigators will collect participant's medication List and Past Medical History.

Then, Investigators would like to ask participants to carry special device on their mid-thigh. It's called 'ActivPAL' and a trained research assistant will fit it on participant's dominant leg. This device has ability to detect the joint angle of participant's thigh to capture lying, sitting, standing, and stepping activities.

Then Investigators will proceed to ultrasound test. Participants will be asked to lay down on the bed with their legs supported by a pillow. Then a study physician will use ultrasound to measure participant's leg muscles. Three measurements will be taken for each participant.

After that participant will be asked to do a "Grip test". Participant will be asked to squeeze special device, called dynamometer, using your dominant hand. Each participant will be asked to make three attempts with half a minute break between each measurement.

Participant will be asked to walk 10-15 meters in order to measure their gait speed.

Impedance measures of body composition will be performed using an automatic scale.

At the end Investigators will ask you to measure participant's body structure, using skinfold/caliper device.

At participant discharge Investigators will remove 'ActivPal' sensor from their leg that was fitted at enrollment.

ELIGIBILITY:
Inclusion Criteria:

* be 65 years of age or older
* be admitted in ACE Unit

Exclusion Criteria:

* be less than 65 years of age
* be nonambulatory
* be diagnosed with end-stage organ failure (end-stage COPD, renal failure requiring dialysis, end-stage heart failure)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Study population will be recruited consecutively from the Acute Care of the Elderly Unit at SPH.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Total standing time | 2 weeks or shorter
  Total upright time will show a strong association with both continuous measures of frailty (Clinical Frailty Scale) and the presence of sarcopenia, as measured by ultrasound and bioelectric impedance measures.

SECONDARY OUTCOMES:
Daily step counts | 2 weeks or shorter
  2. Daily step counts will show strong correlations with patient outcomes (length of stay, readmission rates, discharge to care facility, functional outcomes at 1year, and mortality rates).

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Madden, MD, Principal Investigator — UBC
Locations (1):
- Gerontology Research Lab, Dept. of Medicine, Vancouver Coastal Health Research Institute, VGH Research Pavilion, Room 186-828 West 10th Avenue, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No